CLINICAL TRIAL: NCT03901248
Title: Study of Association of Salivary Adipokines With Prediabetes and Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: IDRFARH005
Record Dates: First submitted 2018-06-04; First posted 2019-04-03 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normoglycemia: Participant with normal blood glucose level with No Intervention
  Interventions: Other: No Intervention
- Impaired Glucose Tolerance: Participants with Impaired Glucose Tolerance blood glucose level with No Intervention
  Interventions: Other: No Intervention
- Type 2 Diabetes: Newly diagnosed type 2 diabetes patients with No Intervention
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Observational study

SUMMARY:
India has more than 65 million adults with Type 2 Diabetes Mellitus (T2DM) and also has a large number with subclinical stages of glycaemia including impaired fasting glucose (IFG) and impaired glucose tolerance (IGT). At present people with high risk of diabetes are identified by blood test such as Oral glucose tolerance Test and/or glycosylated haemoglobin A1c (HbA1c). Dysregulated actions of adipokines have major roles in development of metabolic diseases such as diabetes. Adipokines influence systemic insulin resistance and also regulate inflammatory process and/or are likely to have major pathological role in the development of diabetes. It is also likely that these abnormalities occur even in sub clinical stages of T2DM which when identified would provide an early opportunity to institute early intervention using life style changes which are proven to be effective in all ethnic groups.The measurements of adipokines such as adiponectin, apelin, visfatin and vaspin which have inter related regulatory roles, in saliva if found to be sensitive would provide a non-invasive, simple method of assessing persons with high risk of T2DM.

DETAILED DESCRIPTION:
This study is conducted in a tertiary care hospital, Dr.A.Ramachandran's Diabetes Hospitals, Chennai. The persons with no history of diabetes, seeking a screening for diabetes will be invited to participate in the study and after signing the informed consent form they will be assessed by the risk score. The patients who fulfill the inclusion criteria will be enrolled in this study and additional tests will be done. We will also invite the patient's spouse, relatives or friends who are willing to participant in this study.

Preliminary screening: The team comprises of one research associate (dentist), one research associate, two laboratory technicians and one lab assistant. The measurements will be assessed by the same members of the team throughout screening, to eliminate potential inter-observer variation. Participants aged ≥35 years who visit the clinic will be invited to undergo a preliminary screening. Weight and height are measured with the participants wearing light clothes without shoes. BMI is calculated (kg/m2). Waist circumference is measured midway between the lower rib margin and the iliac crest. Blood pressure is measured using a standard mercury sphygmomanometer after a 5-minute rest. An average of the two readings is used for the analysis. Previous history of hypertension, borderline diabetes and gestational diabetes will be ascertained. Family history of diabetes, heart disease, stroke and sedentary life style are recorded in a structured questionnaire. If the participant has 2 or more risk factors they will be tested for fasting and 2h plasma glucose after 75gm of Oral Glucose (Accu check performa, Roche Diagnostics).

Next day participants will be categorized based on the inclusion and exclusion criteria as Normoglycemic, Pre diabetic (IFG/IGT) and newly diagnosed Type 2 diabetic patients. The selected participants will undergo dental examination to check for periodontitis. Then salivary and fasting serum sample is obtained from all the individuals for estimation of biomarkers (adiponectin, apelin, visfatin and vaspin). HbA1c, Lipid profile and Gamma-glutamyl transferase (GGT) is analysed in fasting serum.

Approximately 10 ml blood is collected in a serum tube. Blood sample separation is performed at the central investigational laboratory. Blood samples are separated, aliquoted, refrigerated and immediately stored at -70˚C for biomarker analysis. HbA1c is measured by immunoturbidometry (tina-quant II; roche diagnostics corporation, germany); a procedure certified by the national glycohemoglobin standardization programme. The fasting serum lipid profile (total cholesterol, triglycerides and high density lipoprotein, cholesterol) and GGT is estimated using standard enzymatic methods. Biochemical assays are performed on a Cobas Integra 450 plus (Roche, Germany) autoanalyzer using reagents from Roche diagnostics, with appropriate quality control methods (Roche diagnostics reference serum).

Unstimulated salivary samples will be collected in a sample collection tube. Participant will be asked to refrain from eating or drinking for about two hours prior to saliva collection; it is done around 8am - 10am. Subjects will be asked to rinse their mouth with drinking water and then to expectorate whole saliva in a collection tube. The saliva is then centrifuged at 9300g at 40 C for about 10 minutes and then stored at -70 degree C, until further use.

Saliva and plasma will be thawed at room temperature for biomarkers measurement by enzyme-linked immunosorbent assay (ELISA). A commercial ELISA kit for human biomarkers for serum and saliva is used and the assay is conducted according to the manufacturer's instructions. Each sample of saliva and plasma from the same patient will be analysed in the same experimental set. Plasma samples require dilution. Saliva samples will be analyzed without dilution.

Reports will be dispatched from the central laboratory to the participants by courier. Participants with newly diagnosed diabetes or uncontrolled diabetes will be referred to a diabetologist for treatment and followed up for two year. Individuals with prediabetes will be advised to improve physical activity and dietary habits and followed up for two year. Participants with periodontitis will be referred to a dental surgeon and followed up for two year.

During visit 4 & 6 the participant's weight, waist circumference, BMI, blood pressure will be measured and laboratory investigations like Fasting and 2hr postprandial blood glucose, HbA1c and Lipid profile. At Visit 6 the participant's saliva and serum samples are collected for adipokines measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Particpants both men and women will be selected for screening using risk factors for diabetes such as age ≥ 35 years, family history of diabetes, previous history of hypertension, sedentary life-style, gestational diabetes, previous history of borderline diabetes, waist circumference ≥ 90 cm males & ≥ 80cm in females, Body Mass Index (BMI) ≥ 23kg/m2. 2hr plasma glucose will be done for those subjects who have 3 or more risk factors.
2. Arm 1: 2hr plasma glucose after 75gm of Glucose - < 140 mg/dl
3. Arm 2: 2hr plasma glucose after 75gm of Glucose - ≥ 140 mg/dl to < 199 mg/dl
4. Arm 3: 2hr plasma glucose after 75gm of Glucose - ≥ 200 mg/dl
5. Have given written informed consent to participate in this study in accordance with local regulations

Exclusion Criteria:

1. Smokers for over a period of 6 months (1 or more cigarettes per day).
2. Beetle nut chewer over a period of 3 months.
3. Patients with bleeding disorders
4. Patients who require antibiotic prophylaxis prior to dental treatment.
5. History of antibiotic therapy within 3 months prior to the study
6. Patients with uncontrolled systemic disease
7. Partipants who is not willing to participate in the study
8. Individuals who are cognitively impaired and/or who are unable to give informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normoglycemic, prediabetic and newly diagnosed Type 2 diabetic participants
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Interrelationship of adipokines such as adiponectin, apelin, visfatin and vaspin in different glycaemic stages | Baseline and 2 years
  Levels of adiponectin, visfatin, vaspin and apelin in prediabetes and diabetes

SECONDARY OUTCOMES:
Change in BMI | Baseline and 2 years
  BMI changes
Change in Blood Pressure | Baseline and 2 years
  Blood Pressure changes
Change in fasting blood glucose | Baseline and 2 years
  Blood pressure Changes
Change in postprandial blood glucose | Baseline and 2 years
  Postprandial blood glucose changes
Comparative assessment of the sensitivity of the assays of the biomarkers in saliva and serum | Baseline and 2 years
  The sensitivity of biomarkers in saliva and serum
Levels of these biomarkers in the presence of periodontitis | Baseline and 2 years
  Relationship of Biomarkers in the presence of periodontitis
Change in HbA1c | Baseline and 2 years
  HbA1c changes

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ramachandran Ambady, MD,PhD,DSc, Study Chair — President, India Diabetes Research Foundation

IPD SHARING:
Plan to Share IPD: Undecided